CLINICAL TRIAL: NCT00189488
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate Palifermin (rHuKGF) in the Reduction of Acute Graft Versus Host Disease in Subjects With Hematologic Malignancies Undergoing Allogeneic Marrow/PBPC Transplantation
Brief Title: Trial to Evaluate Palifermin in the Reduction of Acute Graft Versus Host Disease in Patients With Hematologic Malignancies Undergoing Allogeneic Marrow/Peripheral Blood Progenitor Cell (PBPC) Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20040213; NCT00964899 (obsolete NCT alias)
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Graft Versus Host Disease; Hematologic Malignancies
Keywords: Hematological Malignancies; Graft-versus-host-disease; Oral Mucositis; Allogeneic Transplantation
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms; Stomatitis | interventions — Fibroblast Growth Factor 7; Transplantation Conditioning; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Palifermin (Experimental): Palifermin 60 μg/kg administered daily on 3 consecutive days prior to the day of start of the conditioning regimen and 180 μg/kg administered once prior to transplant and at least 96 hours from last palifermin dose of 60 μg/kg. Participants received conditioning therapy starting at least 24 hours after the last 60 μg dose of palifermin. Allogeneic stem cell transplant occurred on Day 0. Methotrexate dosing began at least 24 hours after the 180 μg/kg dose of palifermin on Days 1, 3, 6 and (planned) 11 administration (toxicity allowing) at doses of 15, 10, 10 and 10 mg/m^2 respectively.
  Interventions: Drug: Palifermin; Other: Conditioning Regimen; Procedure: Allogeneic stem cell transplant; Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo to palifermin 60 μg/kg administered daily on 3 consecutive days prior to the day of start of the conditioning regimen and placebo to palifermin 180 μg/kg once prior to transplant and at least 96 hours from previous placebo to palifermin 60 μg/kg dose. Participants received conditioning therapy starting at least 24 hours after the last 60 μg/kg dose of placebo to palifermin. Allogeneic stem cell transplant occurred on Day 0. Methotrexate dosing began at least 24 hours after the dose of placebo to palifermin 180 μg/kg on Days 1, 3, 6 and (planned) 11 administration (toxicity allowing) at doses of 15, 10, 10 and 10 mg/m^2 respectively.
  Interventions: Drug: Placebo; Other: Conditioning Regimen; Procedure: Allogeneic stem cell transplant; Drug: Methotrexate

INTERVENTIONS:
Drug: Palifermin — Administered as an intravenous (IV) bolus.
  Other Names: Recombinant human keratinocyte growth factor (rHuKGF); Kepivance
  Arms: Palifermin
Drug: Placebo — Administered as an intravenous (IV) bolus.
  Arms: Placebo
Other: Conditioning Regimen — Each participant received 1 of the following conditioning regimens:
  * Cyclophosphamide (Cy) / total body irradiation (TBI) with and without etoposide (VP-16)
  * TBI/VP-16
  * Melphalan (Mel)/TBI (TBI regimens must include fully ablative doses ie > 1100 cGy; sequence of chemotherapy/radiation (CT/RT) flexible)
  * Busulfan (Bu)/Cy
  * Bu/Mel (non-TBI but fully ablative regimens/doses [Mel dose > 140 mg/m^2])
  * Fludarabine (Flu)/Mel (non-TBI but fully ablative regimens/doses [Mel dose > 140 mg/m^2])
Procedure: Allogeneic stem cell transplant — Allogeneic marrow/peripheral blood progenitor cell transplantation
Drug: Methotrexate

SUMMARY:
The main purpose of this study is to evaluate the effect of palifermin versus placebo in the reduction of severe acute graft versus host disease (GVHD) and severe oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hematologic malignancies (including myelodysplastic syndromes [MDS]) who are considered eligible for Cyclophosphamide (Cy)/Total Body Irradiation(TBI) +/- Etoposide (VP-16); Total Body Irradiation(TBI)/ Etoposide(VP-16); Melphalan(Mel) / Total Body Irradiation(TBI); Busulfan(Bu)/ Cyclophosphamide(Cy); Busulfan(Bu)/ Melphalan (Mel); or Fludarabine(Flu)/ Melphalan(Mel) conditioning therapy with allogeneic stem cell support
* Subjects with a 6/6 Human Leukocyte Antigen (HLA)-matched family member or unrelated donor who would provide donor marrow/ peripheral progenitor stem cells. [For unrelated matched donors, molecular typing of class I and class II is mandatory]
* Karnofsky Performance Status >= 70%
* 18 years of age or older at time of informed consent
* Before any study-specific procedure, the appropriate written informed consent must be obtained

Exclusion Criteria:

* Cancer other than Non-Hodgkin's lymphoma, Hodgkin's disease, acute myelogenous leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic lymphocytic leukemia, myelodysplastic syndrome or multiple myeloma (except: adequately treated basal cell carcinoma of the skin)
* Prior autologous or allogeneic bone marrow or peripheral blood stem cell transplantation
* Previous use of palifermin
* Current active infection (including human immunodeficiency virus (HIV) and hepatitis) or oral mucositis
* Congestive heart failure as defined by New York Heart Association class III or IV
* Graft T-cell depletion for Graft-versus-host disease (GVHD) prophylaxis
* Inadequate renal function (serum creatinine > 1.5x the upper limit of normal per the institutional guidelines or clearance < 40 ml/min adjusted for age)
* Inadequate liver function (total bilirubin > 1.5x the upper limit of normal, aspartate aminotransferase (AST) > 3x upper limit of normal and/or alanine aminotransferase (ALT) > 3x upper limit of normal per the institutional guidelines)
* Inadequate pulmonary function as measured by a corrected DLCO (diffusing capacity of the lung for carbon monoxide lung function test) <50% of predicted
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)
* Subject of child-bearing potential is evidently pregnant (e.g. positive human chorionic gonadotropin- HCG test) or is breast feeding during Part A of the study
* Subject or partner of subject is not using or refuses to use adequate contraceptive precautions during Part A of the study
* Subject has known sensitivity to any of the products to be administered during dosing including Escherichia coli-derived products
* Subject was previously randomized into this study
* Subject will not be available for follow-up assessments
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-12; Primary Completion 2008-11 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo to 60 μg/kg palifermin administered daily on 3 consecutive days prior to the day of start of the conditioning regimen and placebo to 180 μg/kg palifermin once prior to transplant and at least 96 hours from the previous placebo dose. Participants received conditioning therapy starting at least 24 hours after the last 60 μg/kg dose of placebo to palifermin. Allogeneic stem cell transplant occurred on Day 0. Methotrexate dosing began at least 24 hours after the dose of placebo to palifermin 180 μg/kg on Days 1, 3, 6 and (planned) 11 administration (toxicity allowing) at doses of 15, 10, 10 and 10 mg/m^2 respectively.
Period: Overall Study
Arm/Group | Placebo | Palifermin
Started | 78 | 77
Received Palifermin/Placebo | 75 | 76
Completed | 63 | 55
Not Completed | 15 | 22
Not completed — Ineligibility determined | 1 | 0
Not completed — Protocol deviation | 2 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Disease progression | 2 | 4
Not completed — Administrative Decision | 0 | 2
Not completed — Death | 5 | 8
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo to 60 μg/kg palifermin administered daily on 3 consecutive days prior to the day of start of the conditioning regimen and placebo to 180 μg/kg palifermin administered once, prior to transplant and at least 96 hours from the previous placebo dose.
- Palifermin: Palifermin 60 μg/kg administered daily on 3 consecutive days prior to the day of start of the conditioning regimen and 180 μg/kg administered once prior to transplant and at least 96 hours from last palifermin dose of 60 μg/kg.
- Total: Total of all reporting groups
Arm/Group | Placebo | Palifermin | Total
Number analyzed (Participants) | 78 | 77 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (10.5) | 40.4 (12.1) | 41.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 37 | 66
  Male | 49 | 40 | 89
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 67 | 65 | 132
  Black or African American | 4 | 3 | 7
  Hispanic or Latino | 4 | 5 | 9
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 0 | 1 | 1
Type of diagnosis [Number; unit: participants] — Acute lymphoblastic leukemia, acute myelogenous leukemia, chronic lymphocytic leukemia, and chronic myelogenous leukemia are subsets of leukemia.
  participants
    Leukemia - all types | 62 | 55 | 117
    Acute lymphoblastic leukemia | 15 | 17 | 32
    Acute myelogenous leukemia | 34 | 29 | 63
    Chronic lymphocytic leukemia | 7 | 3 | 10
    Chronic myelogenous leukemia | 6 | 6 | 12
    Hodgkin's disease | 0 | 1 | 1
    Non-Hodgkin's lymphoma | 6 | 9 | 15
    Multiple Myeloma | 1 | 0 | 1
    Myelodysplastic Syndrome | 9 | 12 | 21
Donor type [Number; unit: participants]
  Related Family Member | 46 | 45 | 91
  Unrelated | 32 | 32 | 64
Donor source [Number; unit: participants]
  Marrow | 17 | 18 | 35
  Peripheral blood progenitor cell(s) | 61 | 59 | 120
Prior radiotherapy [Number; unit: participants]
  Yes | 3 | 4 | 7
  No | 75 | 73 | 148

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Grade 2 to 4 Acute Graft Versus Host Disease (GVHD)
Description: GVHD was graded using the modified Keystone Criteria weekly during the first 2 months after stem cell infusion, then every other week until Day 100.
  Severity was determined clinically (based on physical exam and laboratory serum values) and from biopsies of affected organs whenever possible. The degree of GVHD in individual organs was scored by at least 2 assessors.
  Grade 2 GVHD = > 50% skin involvement or total bilirubin 2.0 - 3.0 mg/dL or 500 - 999 mL/day diarrhea, or persistent nausea with histologic evidence.
  Grade 3 GVHD = total bilirubin 3.1 - 15.0 mg/dL or ≥ 1000 mL/day diarrhea or severe abdominal pain with/without ileus.
  Grade 4 GVHD = skin involvement with bullous formation or total bilirubin > 15.0 mg/dL.
Time Frame: From transplant (Day 0) until Day 100
Population: Primary Analysis Set (consisting of all randomized participants) with GVHD assessments.
Measure: Number; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 72 | 74
Participants
  Yes | 29 | 43
  No | 43 | 31
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel; Adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights; Adjusted Treatment Difference (%) = -17.9, 95% CI 2-sided [-33.4 to -2.4] — The difference between treatment groups in the percentage of participants with Grade 2 to 4 acute GVHD, adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights

2. Primary Outcome: Number of Participants With Severe (Grade 3 and 4) Acute Graft Versus Host Disease (GVHD)
Description: GVHD was graded using the modified Keystone Criteria weekly during the first 2 months after stem cell infusion, then every other week until Day 100.
  Severity was determined clinically (based on physical exam and laboratory serum values) and from biopsies of affected organs whenever possible. The degree of GVHD in individual organs was scored by at least 2 assessors.
  Grade 3 GVHD = total bilirubin 3.1 - 15.0 mg/dL or ≥ 1000 mL/day diarrhea or severe abdominal pain with/without ileus.
  Grade 4 GVHD = skin involvement with bullous formation or total bilirubin > 15.0 mg/dL.
Time Frame: From transplant (Day 0) until Day 100
Population: Primary Analysis Set (consisting of all randomized participants) with GVHD assessments. Efficacy analyses were according to randomized treatment assignment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 72 | 74
Participants
  Yes | 12 | 12
  No | 60 | 62
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.929, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Difference (%) = 0.5, 95% CI 2-sided [-11.0 to 12.1] — The difference between treatment groups in the percentage of participants with severe GVHD, adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights

3. Secondary Outcome: Number of Participants With Day 11 Methotrexate Graft Versus Host Disease Prophylaxis Administration
Description: Low dose methotrexate is widely used in regimens to prophylax against acute GVHD. Methotrexate was administered on days 1, 3, 6 and 11 (toxicity allowing) at doses of 15, 10, 10 and 10 mg/m^2, respectively.
Time Frame: Day 11
Population: Primary Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 78 | 77
Participants
  Yes | 56 | 60
  No | 22 | 17
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.352, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference (%) = -6.5, 95% CI 2-sided [-19.4 to 6.4] — The difference between treatment groups in the percentage of participants with Day 11 Methotrexate GVHD, adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights

4. Secondary Outcome: Number of Participants With Severe (Grade 3 or 4) Oral Mucositis
Description: Oral cavity assessments were performed by a trained assessor using the World Health Organization (WHO) oral toxicity scale. Daily oral mucositis assessments were performed:
  * while participants were hospitalized, including the day of discharge (maximum until day 28);
  * after discharge until the oral mucositis grade returns to a WHO grade ≤ 2.
  The WHO oral toxicity criteria are: Grade 0 = None; Grade 1 = Soreness, erythema; Grade 2 = Erythema, ulcers, ability to eat solids; Grade 3 = Ulcers, requires liquid diet; Grade 4 = Alimentation not possible.
Time Frame: From transplant (Day 0) until Day 100
Population: Primary Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 78 | 77
Participants
  Yes | 57 | 62
  No | 16 | 13
  Unknown | 5 | 2
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Participants with "Unknown" incidence are treated as "Yes" when constructing the differences, 95% confidence intervals and p-value; Test type: Superiority or Other; p = 0.675, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference (%) = -2.6, 95% CI 2-sided [-14.2 to 9.0] — Difference between treatment groups in the percentage of participants with severe oral mucositis, adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights

5. Secondary Outcome: Duration of Severe Oral Mucositis (WHO Grade 3 and 4)
Description: The duration of severe oral mucositis was calculated as the number of days from the onset of severe mucositis (first time a WHO grade of 3 or 4 was observed) to the last day when severe mucositis was observed. If oral mucositis assessments were recorded as missed visits immediately prior to or immediately after severe mucositis was recorded, the missed visits were considered to be severe oral mucositis.
Time Frame: From transplant (Day 0) until Day 100
Population: Primary Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 78 | 77
days | 8.1 (6.8) | 7.8 (6.7)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.953, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 0.5, 95% CI 2-sided [-1.5 to 2.5] — Adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights

6. Secondary Outcome: Number of Participants With Parenteral or Transdermal Opioid Analgesic Use
Description: Includes nonprophylactic intravenous opioid analgesics (fentanyl, morphine, morphine sulphate, hydromorphone, meperidine) and transdermal opioid analgesics (fentanyl patch) for the indication of oral mucositis and dysphagia.
Time Frame: From transplant (Day 0) until Day 100
Population: Primary Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 78 | 77
Participants
  Yes | 50 | 48
  No | 28 | 29
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.797, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference (%) = 2.0, 95% CI 2-sided [-12.5 to 16.5] — Difference between treatment groups in the percentage of participants with opioid analgesic use, adjusted for the stratification factors (TBI use, matched donor type, and source of donor cells) using the Cochran-Mantel-Haenszel weights

7. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization was defined as the number of days a participant stayed in hospital (hospitalized) during the period starting from the day of the transplant (Day 0) to the 100th day following the transplant.
Time Frame: From transplant (Day 0) until Day 100
Population: Primary analysis set
Measure: Mean (Standard Deviation); unit: days
Groups:
- Palifermin: PaPalifermin 60 μg/kg administered daily on 3 consecutive days prior to the day of start of the conditioning regimen and 180 μg/kg administered once prior to transplant and at least 96 hours from last palifermin dose of 60 μg/kg.
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 78 | 77
days | 36.1 (20.8) | 42.2 (25.1)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.186, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = -5.5, 95% CI 2-sided [-12.7 to 1.8] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Area Under the Curve (AUC) of Mouth and Throat Soreness Score
Description: The modified Oral Mucositis Daily Questionnaire (OMDQ) is a self-reported tool that evaluates overall health, mouth and throat soreness (MTS) and activity limitations due to MTS.
  The modified OMDQ was completed once daily beginning with the first day of study drug administration through day 28.
  The area under the curve of mouth and throat soreness score was assessed from the question "How much mouth and throat soreness did you experience in the past 24 hours?" Participants answered on a scale from 0 (no soreness) to 4 (extreme soreness).
Time Frame: The first day of study drug administration through Day 28.
Population: Primary analysis set
Measure: Mean (Standard Deviation); unit: MTS score * days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 78 | 77
MTS score * days | 43.0 (26.3) | 47.7 (26.2)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.219, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = -4.1, 05% CI 2-sided [-12.2 to 4.0] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: 125 Days
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Two participants were randomized to the Placebo arm but received palifermin inadvertently and were summarized in Palifermin arm.
Arm/Group | Placebo | Palifermin
Serious Adverse Events (participants affected / at risk) | 40/73 | 50/78
Other Adverse Events (participants affected / at risk) | 71/73 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Palifermin (N=78)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Caecitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 10 | 10
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Graft versus host disease (Immune system disorders) | 12 | 17
Graft versus host disease in liver (Immune system disorders) | 0 | 1
Immunodeficiency (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 1
Bacteraemia (Infections and infestations) | 5 | 2
Bacterial infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 2
Catheter sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 1
Enterobacter infection (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 2 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Mycobacterial infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia aspergillus (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 5
Septic shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 3 | 4
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Medical device pain (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Atrial natriuretic peptide increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood culture (Investigations) | 0 | 1
Cytomegalovirus antigen positive (Investigations) | 1 | 0
Cytomegalovirus test (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Oral intake reduced (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Unresponsive to verbal stimuli (Nervous system disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cryptogenic organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Venoocclusive disease (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Palifermin (N=78)
Anaemia (Blood and lymphatic system disorders) | 14 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 24 | 24
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Pancytopenia (Blood and lymphatic system disorders) | 5 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 13
Bradycardia (Cardiac disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 16 | 20
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Cushingoid (Endocrine disorders) | 4 | 2
Conjunctival haemorrhage (Eye disorders) | 1 | 4
Dry eye (Eye disorders) | 5 | 5
Vision blurred (Eye disorders) | 9 | 9
Abdominal discomfort (Gastrointestinal disorders) | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 10
Abdominal pain (Gastrointestinal disorders) | 27 | 34
Abdominal pain upper (Gastrointestinal disorders) | 4 | 6
Abdominal tenderness (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 29 | 16
Diarrhoea (Gastrointestinal disorders) | 65 | 64
Dry mouth (Gastrointestinal disorders) | 13 | 11
Dyspepsia (Gastrointestinal disorders) | 12 | 16
Dysphagia (Gastrointestinal disorders) | 10 | 6
Flatulence (Gastrointestinal disorders) | 6 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 3
Haemorrhoids (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 70 | 71
Oesophagitis (Gastrointestinal disorders) | 2 | 7
Oral pain (Gastrointestinal disorders) | 6 | 9
Paraesthesia oral (Gastrointestinal disorders) | 1 | 4
Proctalgia (Gastrointestinal disorders) | 7 | 4
Tongue coated (Gastrointestinal disorders) | 2 | 7
Tongue disorder (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 53 | 53
Asthenia (General disorders) | 18 | 15
Catheter site pain (General disorders) | 9 | 8
Chills (General disorders) | 13 | 7
Face oedema (General disorders) | 3 | 6
Fatigue (General disorders) | 47 | 54
Generalised oedema (General disorders) | 2 | 5
Mucosal inflammation (General disorders) | 8 | 12
Oedema (General disorders) | 11 | 9
Oedema peripheral (General disorders) | 30 | 26
Pain (General disorders) | 11 | 6
Pyrexia (General disorders) | 33 | 34
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 4
Jaundice (Hepatobiliary disorders) | 2 | 4
Graft versus host disease (Immune system disorders) | 17 | 13
BK virus infection (Infections and infestations) | 3 | 4
Bacteraemia (Infections and infestations) | 9 | 11
Candidiasis (Infections and infestations) | 2 | 8
Catheter site infection (Infections and infestations) | 4 | 1
Clostridial infection (Infections and infestations) | 4 | 3
Cytomegalovirus viraemia (Infections and infestations) | 2 | 4
Enterococcal infection (Infections and infestations) | 4 | 5
Folliculitis (Infections and infestations) | 5 | 2
Oral candidiasis (Infections and infestations) | 2 | 9
Pneumonia (Infections and infestations) | 1 | 4
Staphylococcal infection (Infections and infestations) | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 8
Contusion (Injury, poisoning and procedural complications) | 5 | 3
Blood bilirubin increased (Investigations) | 0 | 4
Blood creatinine increased (Investigations) | 4 | 1
Cytomegalovirus test (Investigations) | 3 | 6
Weight decreased (Investigations) | 8 | 6
Anorexia (Metabolism and nutrition disorders) | 26 | 26
Decreased appetite (Metabolism and nutrition disorders) | 15 | 12
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Fluid overload (Metabolism and nutrition disorders) | 3 | 5
Fluid retention (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 15
Pain in jaw (Musculoskeletal and connective tissue disorders) | 5 | 3
Shoulder pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Dizziness (Nervous system disorders) | 21 | 14
Dysgeusia (Nervous system disorders) | 8 | 6
Headache (Nervous system disorders) | 38 | 46
Lethargy (Nervous system disorders) | 4 | 4
Neuropathy peripheral (Nervous system disorders) | 6 | 2
Paraesthesia (Nervous system disorders) | 4 | 3
Sinus headache (Nervous system disorders) | 4 | 1
Tremor (Nervous system disorders) | 17 | 10
Anxiety (Psychiatric disorders) | 20 | 18
Confusional state (Psychiatric disorders) | 13 | 6
Depression (Psychiatric disorders) | 11 | 10
Hallucination (Psychiatric disorders) | 8 | 5
Insomnia (Psychiatric disorders) | 29 | 28
Dysuria (Renal and urinary disorders) | 9 | 10
Haematuria (Renal and urinary disorders) | 11 | 12
Pollakiuria (Renal and urinary disorders) | 4 | 3
Renal failure (Renal and urinary disorders) | 6 | 6
Renal failure acute (Renal and urinary disorders) | 1 | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Blister (Skin and subcutaneous tissue disorders) | 4 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 4
Erythema (Skin and subcutaneous tissue disorders) | 17 | 11
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 9 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 20
Rash (Skin and subcutaneous tissue disorders) | 27 | 35
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 4
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 10
Flushing (Vascular disorders) | 5 | 4
Hypertension (Vascular disorders) | 25 | 29
Hypotension (Vascular disorders) | 13 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.